CLINICAL TRIAL: NCT06236984
Title: Retrospective Data Analysis of CKRT Treatments in Adult Mode With multiFiltratePRO
Brief Title: Retrospective Data Analysis of CKRT (Continuous Kidney Replacement Therapy) Treatments in Adult Mode With multiFiltratePRO
Acronym: CKRT-AKI
Status: Completed | Type: Observational
Sponsor: Fresenius Medical Care Deutschland GmbH (Industry)
Collaborators: Metronomia Clinical Research GMBH (Unknown)
Responsible Party: Sponsor
Other Study IDs: CKRT-AKI-01-EU
Record Dates: First submitted 2024-01-05; First posted 2024-02-01 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Acute Kidney Injury; Renal Failure
Keywords: Continuous kidney replacement therapy
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- AKI patients: Patients with an indication for the extracorporeal blood treatment suffering from AKI who received CKRT adult mode treatment
  Interventions: Other: multiFiltratePRO with all CKRT treatment modes

INTERVENTIONS:
Other: multiFiltratePRO with all CKRT treatment modes — Retrospective Data Analysis of CKRT treatments in adult mode with multiFiltratePRO

SUMMARY:
The multiFiltratePRO is a device for extracorporeal blood purification treatments.

In this retrospective analysis, the treatments of patients who received at least one treatment with the investigational device as mentioned between January 2015 and January 2024 will be documented in a chronological order. No further control treatments will be investigated in this one-arm design. The design is considered to be appropriate to reflect daily clinical practice and to contribute to empirical evidence of performance of the multiFiltratePRO system.

ELIGIBILITY:
Inclusion Criteria:

* All patients with an indication for the extracorporeal blood treatment suffering from AKI who received CKRT adult mode treatment for at least once with: Heparin-Continuous veno-venous hemofiltration Hep-CVVH (Pre CVVH, Post CVVH and Pre-Post CVVH), Heparin-Continuous veno-venous hemodialysis Hep-CVVHD, Heparin-Continuous veno-venous hemodiafiltration Hep-CVVHDF (Pre-CVVHDF and Post-CVVHDF), Citrate-Calcium(Ci-Ca)-CVVHD, Citrate-Calcium(Ci-Ca) CVVHDF, between January 2015 and January 2024, with the investigational device, have to be included in the study in chronological order.
* No age restriction for heparin modes
* Age ≥ 18 years for Ci-Ca modes at treatment start
* Patient´s body weight ≥ 40kg irrespective of age
* Acute Kidney Injury (AKI) OR chronic dialysis patients with clinical indication for CKRT

Exclusion Criteria:

* Participation in an interventional clinical study during the retrospectively collected CKRT treatment data
* Previous participation in the same study
* No study-specific exclusion criteria based on contraindications due to the retrospective character of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with an indication for the extracorporeal blood treatment suffering from AKI who received CKRT adult mode treatment
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-02-21 (Actual); Study Completion 2025-02-21 (Actual)

PRIMARY OUTCOMES:
Analysis of treatments with multiFiltratePRO | documentation of max.7 treatment days
  Performance data of defined multiFiltratePRO CKRT treatments in adult mode with regard to fluid balance (effluent dose) are analysed

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Borgstedt, Dr. med., Principal Investigator — Evangelisches Klinikum Bethel gGmbH Universitätsklinikum OWL der Universität Bielefeld
Locations (3):
- Germany (3):
  - Evangelisches Klinikum Bethel gGmbH Universitätsklinikum OWL der Universität Bielefeld, Bielefeld, North Rhine-Westphalia
  - Klinikum Leverkusen gGmbH, Leverkusen, North Rhine-Westphalia
  - Klinikum Ludwigshafen, Ludwigshafen am Rhein, Rhineland-Palatinate

IPD SHARING:
Plan to Share IPD: No